CLINICAL TRIAL: NCT06331338
Title: Research on the Effectiveness of Using Decision Cycle for Person-Centered Glycemic Management on Self-Care Behaviors in Outpatients With Type 2 Diabetes
Brief Title: Effects of Using Decision Cycle for Person-Centered Glycemic Management in Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202310085RIND
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
Keywords: Decision Cycle for Person-Centered Glycemic Management; Self-Care Behaviors; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New health education:use [Decision Cycle for Person-Centered Glycemic Management ] (Experimental): It is a person-centered approach to care. Treatment goals and plans should be cotreated with people with diabetes based on their individual preferences, values, and goals.
  Interventions: Behavioral: Decision Cycle for Person-Centered Glycemic Management
- Traditional diabetes self-management education (Active Comparator): It is a educator-centered approach to care.
  Interventions: Other: Traditional diabetes self-management education

INTERVENTIONS:
Behavioral: Decision Cycle for Person-Centered Glycemic Management — It is defined as a purposefully designed holistic care intervention that improve self-management .
  Arms: New health education:use [Decision Cycle for Person-Centered Glycemic Management ]
Other: Traditional diabetes self-management education — Traditional diabetes self-management education content focuses more on teaching relevant knowledge and some skills.
  Arms: Traditional diabetes self-management education

SUMMARY:
Decision cycle for person-centered glycemic management is a new diabetes decision making .It is defined as a purposefully designed holistic care intervention .The goal is to improve the self-care behavior of patients with type 2 diabetes, thereby improving glycated hemoglobin levels and delaying the occurrence of complications.

DETAILED DESCRIPTION:
The "Decision Cycle for Person-Centered Glycemic management" jointly proposed by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD) in 2018 , which develops treatment goals and plans based on the patient's personal preferences, values, and goals.

Participants will be divided into two groups(treatment group 、control group).Treatment group will accept the "Decision Cycle for Person-Centered Glycemic Management " .It is a person-centered diabetes decision making. Control group will accept the traditional diabetes self-management education. It content focuses more on teaching relevant knowledge and some skills.It is a educator-centered approach.

Baseline / pre-intervention test (after signing informed consent form) post-intervention test (after finishing intervention) Researchers will compare treatment group and control group to see if treatment group has better performance on self-care Behaviors and glycated hemoglobin levels .

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with type 2 diabetes by a physician.
2. Age: 18 years or above.
3. Glycated hemoglobin (HbA1c ) test value: 7.5-9.0 %
4. No diabetic oral medications, insulin and glucagon-like peptide-1 were replaced in the outpatient when the case was admitted.
5. No pregnancy during the study period.
6. After the researcher explains the purpose of the research, the research subjects agree to join this researcher.
7. Those who are conscious and able to take care of themselves.
8. There is no diagnostic certificate from the American Psychiatric Association's Diagnostic Manual of Mental Disorders, Fourth Edition (DSM-IV)of all mental illnesses.
9. Those who can communicate in Mandarin and Taiwanese.

Exclusion Criteria:

1. Patients diagnosed with type 1 diabetes by a physician.
2. Age: Under 18 years old.
3. Glycated hemoglobin test value: less than 7.5 % and greater than 9.0 %
4. Those who replaced oral diabetes medications, insulin and glucagon-like peptide- 1 at the outpatient at the time of admission.
5. Pregnancy during the study period.
6. Those who are unable to take care of themselves and express themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
glycemic control (HbA1c) | Before the task and 3 months post intervention
  The HbA1c level is a marker of the average blood glucose levels over a period of the last 2-3 months.

SECONDARY OUTCOMES:
Diabetes Self-Care Behavior Scale | Before the task and 3 months post intervention
  It is contains 20 likert-scaled (1-5) items, it assessed the frequency with which patients performed the diabetes self-care behaviors, including how often took diabetes medications, exercise, blood glucose monitor, diet . A higher score indicates greater self care behavior .

CONTACTS AND LOCATIONS:
Overall Officials: Kang-Chih Fan, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No